CLINICAL TRIAL: NCT00721565
Title: An Exercise Intervention for Breast Cancer Patients: Feasibility and Effectiveness (BEAT Cancer Trial)
Brief Title: An Exercise Intervention for Breast Cancer Patients: Feasibility and Effectiveness (BEAT Cancer Trial; Pilot Study)
Acronym: BEAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROG-SCCI 08-001-1; SCRIHS 05-071 (Other: Institutional Review Board); E200634 (Other Grant/Funding Number: Excellence in Academic Medicine SIUSM)
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Exercise; Social Cognitive Theory; Adherence; Symptoms; Body Composition
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): behavior change intervention
  Interventions: Behavioral: Exercise Behavior Change
- 2 (No Intervention): written materials

INTERVENTIONS:
Behavioral: Exercise Behavior Change — attend 12 supervised exercise sessions, attend 6 group sessions with psychologist, attend 3 counseling sessions with exercise specialist
  Arms: 1

SUMMARY:
"Translation" of the current "basic science" information related to physical activity into patient intervention programs is needed. This translation is critical to providing benefit to the maximum number of patients. Little is known about the determinants of physical activity among breast cancer patients undergoing hormonal therapy and few studies have attempted to evaluate an exercise behavior change program aimed to improve exercise adherence among such patients. The proposed project will evaluate use of an innovative behavioral and psychosocial intervention to increase physical activity among breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients between the ages of 18 and 70 years of age with a diagnosis of Stage I, II, or IIIA breast cancer who are currently taking aromatase inhibitors or selective estrogen receptor modulators for the next 8 months.
* English speaking
* Medical clearance for participation provided by primary care physicians
* If the patient has undergone a surgical procedure, must be at least 6 weeks post-procedure

Exclusion Criteria:

* Diagnosis of dementia or organic brain syndrome
* Medical, psychological or social characteristic that would interfere with ability to fully participate in program activities and assessments (e.g., psychosis, schizophrenia, etc.)
* Contraindication to participation in a regular physical activity program.
* Metastatic or recurrent disease
* Inability to ambulate
* Engaged in >/= 60 minutes of vigorous physical activity or >/= 150 minutes of moderate plus vigorous physical activity per week during the past month.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-04; Primary Completion 2008-02 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
change in physical activity | 6 months

SECONDARY OUTCOMES:
social cognitive and biopsychosocial outcomes | 3 months
social cognitive and biopsychosocial outcomes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Q. Rogers, MD, MPH, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Background] Rogers LQ, Markwell S, Hopkins-Price P, Vicari S, Courneya KS, Hoelzer K, Verhulst S. Reduced barriers mediated physical activity maintenance among breast cancer survivors. J Sport Exerc Psychol. 2011 Apr;33(2):235-54. doi: 10.1123/jsep.33.2.235. PMID 21558582
- [Background] Rogers LQ, Vicari S, Courneya KS. Lessons learned in the trenches: facilitating exercise adherence among breast cancer survivors in a group setting. Cancer Nurs. 2010 Nov-Dec;33(6):E10-7. doi: 10.1097/NCC.0b013e3181db699d. PMID 20562618
- [Background] Rogers LQ, Hopkins-Price P, Vicari S, Markwell S, Pamenter R, Courneya KS, Hoelzer K, Naritoku C, Edson B, Jones L, Dunnington G, Verhulst S. Physical activity and health outcomes three months after completing a physical activity behavior change intervention: persistent and delayed effects. Cancer Epidemiol Biomarkers Prev. 2009 May;18(5):1410-8. doi: 10.1158/1055-9965.EPI-08-1045. Epub 2009 Apr 21. PMID 19383889
- [Background] Rogers LQ, Hopkins-Price P, Vicari S, Pamenter R, Courneya KS, Markwell S, Verhulst S, Hoelzer K, Naritoku C, Jones L, Dunnington G, Lanzotti V, Wynstra J, Shah L, Edson B, Graff A, Lowy M. A randomized trial to increase physical activity in breast cancer survivors. Med Sci Sports Exerc. 2009 Apr;41(4):935-46. doi: 10.1249/MSS.0b013e31818e0e1b. PMID 19276838
- [Derived] Ehlers DK, Rogers LQ, Courneya KS, Robbs RS, McAuley E. Effects of BEAT Cancer randomized physical activity trial on subjective memory impairments in breast cancer survivors. Psychooncology. 2018 Feb;27(2):687-690. doi: 10.1002/pon.4438. Epub 2017 May 11. No abstract available. PMID 28414894